CLINICAL TRIAL: NCT00942071
Title: A Phase I Study to Assess the Safety and Immunogenicity of a New Influenza Vaccine Candidate MVA-NP+M1 in Healthy Adults
Brief Title: A Study to Assess the Safety and Immunogenicity of a New Influenza Vaccine Candidate MVA-NP+M1 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Flu001
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Influenza
Keywords: Influenza; Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. MVA-NP+M1 ID (Experimental): 12 volunteers to receive MVA-NP+M1 via ID route
  Interventions: Biological: MVA-NP+M1
- 2. MVA-NP+M1 IM (Experimental): 16 volunteers to receive MVA-NP+M1 via IM route
  Interventions: Biological: MVA-NP+M1
- 3. MVA-NP+M1 IM upper age group (Experimental): 30 volunteers to receive MVA-NP+M1 via IM route
  Interventions: Biological: MVA-NP+M1

INTERVENTIONS:
Biological: MVA-NP+M1 — 1. Intradermal injection at 5 x 10^7 pfu at day 0
  Arms: 1. MVA-NP+M1 ID
Biological: MVA-NP+M1 — 2.Intramuscular injection at 5 x 10^7 pfu/ml at day 0. Intramuscular injection at 2.5 x 10^8 pfu/ml at day 0
  Arms: 2. MVA-NP+M1 IM
Biological: MVA-NP+M1 — 3.Intramuscular injection at 1.5 x 10^8 pfu/ml at day 0
  Arms: 3. MVA-NP+M1 IM upper age group

SUMMARY:
This is an open label phase I study, to assess the safety of a novel influenza vaccine, MVA-NP+M1. All volunteers recruited will be healthy. Twelve volunteers will be administered with a single dose of 5 x 10^7 pfu of MVA-NP+M1 via the Intradermal (ID) route (group 1). Sixteen volunteers will receive Intramuscular (IM) MVA-NP+M1. The first 8 volunteers will be administered a single dose of 5 x 10^7 pfu of MVA-NP+M1 followed by a further eight receiving 2.5 x 10^8 pfu of MVA-NP+M1 (group 2). The 3rd group will be split into 3 groups of 10 volunteers in the age ranges 50-59, 60-69 and 70 and above and administered intramuscularly with a single dose of 1.5 x 10^8 pfu of MVA-NP+M1. Safety data will be collected. The secondary aim of this study will be to assess the cellular immune responses generated by each dose.

DETAILED DESCRIPTION:
Antibodies against the external proteins of influenza can prevent the virus from infecting cells and either prevent infection or limit the spread of infection. However the surface proteins are highly variable and there is little antibody cross-reactivity between variants. Once a cell has been infected with the virus, it is then vulnerable to T cell attack resulting in the destruction of infected cells so that no more virus can be produced and the infection is controlled. There is evidence from clinical trials of influenza challenge, and animal models that T cell responses can protect in the absence of antibodies. Additionally, since T cells can recognise the highly conserved internal proteins of influenza, cross-subtype protection can be achieved.

Seasonal influenza infection results in a T cell response to the virus which can protect against subsequent infection. However over the course of a few years these responses decline below protective levels. The new vaccine being tested in this study is designed to boost these T cell responses back to protective levels. Even responses that may be too low to be reliably quantified by currently available assays may still be boosted to high levels by a single dose of recombinant MVA. Since the internal proteins vary little between influenza subtypes, this could result in a 'universal' vaccine against influenza A. If the need to continually reformulate the vaccine in response to mutations in the viral coat proteins can be removed, the universal vaccine could be produced in large amounts and used more widely than the existing seasonal 'flu vaccines, thus protecting the population against currently circulating viruses and new virus types that are at present only found in avian species.

There is very little polymorphism of NP and M1 between influenza A isolates. NP is 92% identical between H3N2 and H1N1 strains, and 91% identical between H3N2 and H5N1 strains. M1 is 95% identical between H3N2 and H1N1 strains, and 93% identical between H3N2 and H5N1 strains. This low level of variation appears to allow strong T cell cross-reactivity.

MVA is a highly attenuated strain of vaccinia virus that is unable to replicate efficiently in human cell lines and most mammalian cells. Viral replication is blocked at a late stage of virion assembly, so, importantly, viral and recombinant protein synthesis is unimpaired. This means that MVA is an efficient single round expression vector, incapable of causing infection in mammals. Replication-deficient recombinant MVA has been seen as an exceptionally safe viral vector. This safety in man is consistent with the avirulence of MVA in animal models, where recombinant MVAs have also been shown to be protectively immunogenic as vaccines against viral diseases and cancer. Importantly for a vaccine which may eventually be used in a large proportion of the population, recombinant MVAs expressing HIV antigens have been shown to be safe and immunogenic in HIV-infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 or over, no upper age limit
* Resident in or near Oxford for the duration of the vaccination study
* Able and willing (in the Investigators' opinions) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females, a negative pregnancy test on the day of vaccination and agreement to practice effective contraception for the duration of the study.
* Agreement to refrain from blood donation during the course of the study
* Written informed consent

Exclusion Criteria:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of a recombinant MVA vaccine
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Any history of anaphylaxis in reaction to vaccination
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any chronic illness requiring ongoing or awaiting hospital specialist supervision, other than minor surgical procedures and follow up of surgery over 6 months prior to screening.
* Suspected or known current injecting drug or alcohol abuse (as defined by an alcohol intake of greater than 42 units every week)
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* For females, pregnancy, lactation or willingness/intention to become pregnant during the study
* Any other significant disease, disorder or finding, which, in the opinion of the Investigators, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study.
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis, as determined by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety of a new influenza vaccine, MVA-NP+M1, when administered to healthy volunteers. | 24 months

SECONDARY OUTCOMES:
To assess the cellular immune response generated by a new influenza vaccine, MVA-NP+M1, when administered as a single dose to healthy volunteers. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, D.Phil FRCP, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Churchill Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Ferrara F, Del Rosario JMM, da Costa KAS, Kinsley R, Scott S, Fereidouni S, Thompson C, Kellam P, Gilbert S, Carnell G, Temperton N. Development of Lentiviral Vectors Pseudotyped With Influenza B Hemagglutinins: Application in Vaccine Immunogenicity, mAb Potency, and Sero-Surveillance Studies. Front Immunol. 2021 May 24;12:661379. doi: 10.3389/fimmu.2021.661379. eCollection 2021. PMID 34108964
- [Derived] Antrobus RD, Lillie PJ, Berthoud TK, Spencer AJ, McLaren JE, Ladell K, Lambe T, Milicic A, Price DA, Hill AV, Gilbert SC. A T cell-inducing influenza vaccine for the elderly: safety and immunogenicity of MVA-NP+M1 in adults aged over 50 years. PLoS One. 2012;7(10):e48322. doi: 10.1371/journal.pone.0048322. Epub 2012 Oct 31. PMID 23118984